CLINICAL TRIAL: NCT00807846
Title: A Phase 4, 6-week, Randomized Double Blind, Multicenter, Active-controlled Trial To Evaluate The Effects Of Celecoxib (Celebrex) Or Naproxen On Blood Pressure In Pediatric Subjects With Juvenile Idiopathic Arthritis.
Brief Title: A Study To Evaluate The Effects Of Celecoxib (Celebrex®) Or Naproxen On Blood Pressure In Pediatric Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3191342
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Juvenile Arthritis; Juvenile Rheumatoid Arthritis;Blood Pressure;Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Celecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Experimental)
  Interventions: Drug: Celecoxib
- Naproxen (Experimental)
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 50 mg or 100 mg PO BID for 6 weeks
  Arms: Celecoxib
Drug: Naproxen — Naproxen 7.5 mg/kg PO BID [maximum of 500 mg BID] for 6 weeks
  Arms: Naproxen

SUMMARY:
This Is A Multicenter, Active-Controlled Trial To Evaluate The Effects Of Celecoxib (Celebrex®) Or Naproxen On Blood Pressure In Pediatric Subjects With Juvenile Idiopathic Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Polyarticular (both rheumatoid factor positive and rheumatoid factor negative),oligoarticular and extended oligoarticular JIA for ≥3 months meeting the International League of Associations for Rheumatology (ILAR) criteria for Juvenile Idiopathic Arthritis (JIA)
* Subjects with Systemic JIA with active arthritis in at least 1 joint but without active systemic features are eligible
* ≥2 years of age and <18 years of age prior to the Baseline visit
* Body weight ≥10 kg at the Baseline visit
* Candidate for chronic NSAID therapy in the Investigator's judgment

Exclusion Criteria:

* Psoriatic arthritis, enthesitis-related arthritis, and undifferentiated arthritis types of JIA
* Active systemic features over the prior 12 weeks in children with systemic Juvenile Idiopathic Arthritis (JIA)
* Subjects with psoriatic arthritis, enthesitis-related arthritis, and undifferentiated arthritis should be excluded
* Subjects with active Systemic JIA should not be enrolled

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (18):
  - Catalina Pointe Clinical Research, Inc., Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital-San Diego, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center / Division of Rheumatology, Washington D.C., District of Columbia
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - Delray Research Associates, Delray Beach, Florida
  - Miami Children's Hospital, Miami, Florida
  - Administrative Site-Hawaii Pacific Health Research Institute, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kosair Charities Pediatric Clinical Research Unit - University of Louisville, Louisville, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University Pediatric Rheumatology of Kentucky, Louisville, Kentucky
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center Pediatric Research Office, Omaha, Nebraska
  - Akron Children's Hospital, Akron, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
- Chile (2):
  - Hospital Regional de Concepcion Guillermo Grant Benavente, Concepción, Región del Biobío
  - Hospital Roberto del Rio, Santiago, RM
- Instituto de Atencion Pediatrica, San José, Costa Rica
- Peru (2):
  - Clinica San Borja/Centro de Investigacion de Reumatologia, San Borja, Lima region
  - Clinica Ricardo Palma/Sitio de Investigacion de Reumatologia, San Isidro, Lima region
- Philippines (2):
  - Philippine General Hospital, Manila
  - University of Santo Tomas Hospital, Manila
- Russia (4):
  - State Healthcare Institution of Moscow "Izmailovskaya City Children's Hospital", Moscow
  - First Moscow State Medical University I.M. Sechenov of the Minzdravsocrazvitiya of Russia, Moscow
  - Smolensk Regional Clinical Hospital, Smolensk
  - SEIHPE "Smolensk State Medical Academy"of the Minzdravsocrazvitiya of Russia, Smolensk
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Children's Clinic of Internal Medicine, Niš
- Clinical Research Unit, Pretoria, Gauteng, South Africa
- Switzerland (2):
  - CHUV - Unit of Immuno-Allergology and Rhumatology, Ch-1011 Lausanne
  - Universitaets-Kinderspital, Ch-8032 Zuerich
- Ukraine (5):
  - Department of Cardioreumatology, Kharkiv
  - Institute of Pediatrics, Obstetrics and Gynecology, Kiev
  - Kyiv City Children Clinical Hospital #1, Kyiv
  - Crimean State Medical University, Chair of Pediatrics with a course of Children Infectious Diseases, Simferopol
  - Zaporizhzhya Regional Clinical Pediatric Hospital, Zaporizhzhya

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191342&StudyName=A%20Study%20To%20Evaluate%20The%20Effects%20Of%20Celecoxib%20%28Celebrex%AE%29%20Or%20Naproxen%20On%20Blood%20Pressure%20In%20Pediatric%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 4, 6-week, randomized double-blind, multicenter, active-controlled trial in participants with juvenile idiopathic arthritis (JIA). A total of 221 participants were screened into the study in 32 investigator sites.
Pre-assignment Details: A total of 101 participants were randomized to treatment with Celecoxib and 100 participants to treatment with Naproxen. Of these randomized, 100 participants received treatment with Celecoxib and 98 participants received treatment with Naproxen. Three participants were randomized but did not receive any treatment.
Groups:
- Celecoxib: Participants received celecoxib capsules 50 mg twice daily (BID) or 100 mg BID for 6 weeks. The volume/dose of the study medications was determined by the subject's weight at Baseline visit
- Naproxen: Participants received naproxen suspension 7.5 mg/kg BID (maximum dose of 500 mg BID) for 6 weeks. The volume/dose of the study medications was determined by the subject's weight at Baseline visit
Period: Overall Study
Arm/Group | Celecoxib | Naproxen
Started | 100 | 98
Completed | 88 | 94
Not Completed | 12 | 4
Not completed — Adverse Event | 5 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Naproxen | Total
Number analyzed (Participants) | 100 | 98 | 198
Age, Customized [Number; unit: Participants]
  >=2 - <8 Years | 22 | 18 | 40
  >=8 - <13 Years | 34 | 47 | 81
  >=13 - <18 Years | 44 | 33 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 64 | 140
  Male | 24 | 34 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 6/Final Visit
Description: Value at 6 weeks minus value at baseline.
Time Frame: 6 Weeks/Final Visit
Population: Safety population included all randomized participants who received at least one dose of study medication. The Safety Analysis set was used to analyze all BP (blood pressure) measurements.
  For early terminations the last observation carried forward (LOCF) was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeter of mercury)
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 100 | 98
mmHg (millimeter of mercury) | 0.366 (0.70) | -0.734 (0.70)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; The primary analysis was based on 90% confidence interval (CI) for the difference across treatment groups (celecoxib - naproxen) in mean change from baseline in SBP. Change from Baseline in BP was analyzed using analysis of covariance (ANCOVA) with model terms for treatment with baseline height, baseline weight, baseline age, and baseline SBP as covariates. No formal hypothesis testing was applied to the primary analysis; Test type: Superiority or Other; p = 0.274, ANCOVA; Mean Difference (Final Values) = 1.100, 90% CI 2-sided [-0.56 to 2.76]

2. Secondary Outcome: Change From Baseline to Week 2 in SBP.
Description: Value at 2 weeks minus value at baseline.
Time Frame: 2 weeks
Population: Safety population included all randomized participants who received at least one dose of study medication. The Safety Analysis set was used to analyze all BP measurements.
  For early terminations the LOCF was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 100 | 98
mmHg | -0.202 (0.53) | -1.290 (0.53)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; For secondary analyses, 95% CIs for the differences across treatment groups (celecoxib - naproxen) in the mean change from baseline were generated. The change from baseline in BP was analyzed using an ANCOVA model with terms for treatment, baseline height, weight, age and baseline BP as covariates. Secondary analyses were conducted using a two-sided test with α=0.05; Test type: Superiority or Other; p = 0.148, ANCOVA; Mean Difference (Final Values) = 1.088, 95% CI 2-sided [-0.39 to 2.57]

3. Secondary Outcome: Change From Baseline in SBP at Week 4.
Description: Value at 4 weeks minus value at baseline.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 100 | 98
mmHg | -0.170 (0.58) | -2.007 (0.58)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; For secondary analyses, 95% CIs for the differences across treatment groups (celecoxib - naproxen) in the mean change from baseline were generated. The change from baseline in blood pressure was analyzed using an ANCOVA model with terms for treatment, baseline height, weight, age and baseline BP as covariates. Secondary analyses were conducted using a two-sided test with α=0.05; Test type: Superiority or Other; p = 0.027, ANCOVA; Mean Difference (Final Values) = 1.837, 95% CI 2-sided [0.21 to 3.46]

4. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Week 2.
Description: Value at 2 weeks minus value at baseline.
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 100 | 98
mmHg | -1.346 (0.52) | -0.139 (0.52)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.106, ANCOVA; Mean Difference (Final Values) = -1.207, 95% CI 2-sided [-2.67 to 0.26]

5. Secondary Outcome: Change From Baseline in DBP at Week 4.
Description: Value at 4 weeks minus value at baseline.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 100 | 98
mmHg | -0.628 (0.54) | -0.848 (0.54)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.776, ANCOVA; Mean Difference (Final Values) = -0.220, 95% CI 2-sided [-1.30 to 1.74]

6. Secondary Outcome: Change From Baseline in DBP at Week 6/Final Visit
Description: Value at 6 weeks/Final Visit minus value at baseline.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 100 | 98
mmHg | -0.535 (0.54) | -0.356 (0.54)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; For secondary analyses, 95% CIs for the differences across treatment groups (celecoxib - naproxen) in the mean change from baseline were generated. The change from baseline in BP was analyzed using an ANCOVA model with terms for treatment, baseline height, weight, age and baseline blood pressure as covariates. Secondary analyses were conducted using a two-sided test with α=0.05; Test type: Superiority or Other; p = 0.815, ANCOVA; Mean Difference (Final Values) = -0.179, 95% CI 2-sided [-1.69 to 1.33]

7. Secondary Outcome: Change From Baseline in Parent's Assessment of Overall Well-being at Week 6/Final Visit.
Description: The parent/legal guardian evaluated the participant's overall well-being at Baseline and at Week 6 (or Final Visit) by placing one vertical line on the visual analog scale (VAS). The VAS ranged from 0 to 100, with 0 being 'very well' and 100 being 'very poor.
Time Frame: 6 weeks
Population: Modified-Intent-to-Treat (MITT) Population included all randomized participants who received at least one dose of study medication and had at least one post-baseline efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: mm (millimeter)
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 98 | 98
mm (millimeter) | -10.581 (2.081) | -13.614 (2.060)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; Change from Baseline to Week 6 was analyzed using ANCOVA model as well with treatment and Baseline value as a covariate. The LS mean change from Baseline was compared between treatment groups and an appropriate p-value and 95% CI for the difference between the two treatment groups was generated. This analysis was conducted using a two-sided test with α=0.05; Test type: Superiority or Other; p = 0.303, ANCOVA; Mean Difference (Final Values) = 3.033, 95% CI 2-sided [-2.76 to 8.82]

8. Secondary Outcome: Number of Participants With >= 30% Improvement in the Parent's Global Assessment of Overall Well-being at Week 6/Final Visit.
Description: as for outcome 7
Time Frame: Week 6/Final Visit
Population: The MITT Population included all randomized participants who received at least one dose of study medication and had at least one post-baseline efficacy measurement.
Measure: Number; unit: Participants
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 98 | 98
Participants | 47 | 54
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; The number of subjects with at least a 30% improvement in Parent/Guardian's Global Assessment of Overall Well-Being was compared between the two treatment groups using a chi-square test. A 95% CI for the difference in incidence between groups was also computed; Test type: Superiority or Other; p = 0.392, Chi-squared; Mean Difference (Final Values) = -0.061, 95% CI 2-sided [-0.202 to 0.079] — Mean Difference (Final Values) indicates difference in incidence (proportion) between treatments

9. Secondary Outcome: Change From Baseline in Participant's Assessment of Overall Well-being at Week 6/Final Visit.
Description: Participants, ≥8 years of age at the baseline, evaluated their own overall well-being at Baseline and at Week 6 (or Final Visit) by placing one vertical line on the VAS. The VAS ranges from 0 to 100, with 0 being 'very well' and 100 being 'very poor'.
Time Frame: 6 weeks
Population: MITT population was used. Additional 3 participants aged <8 yrs at Baseline in Naproxen Arm provided self-assessments. In Celecoxib Arm, 2 participants (>=8 yrs) not provided self-assessment and 2 (>=8 yrs) provided but they were not from MITT and were excluded; additional 1 participant (<8 yrs) provided self-assessment and included in analysis.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 75 | 83
mm | -12.990 (2.226) | -12.588 (2.115)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.897, ANCOVA; Mean Difference (Final Values) = -0.402, 95% CI 2-sided [-6.50 to 5.69]

10. Secondary Outcome: Number of Participants With >= 30% Improvement in the Participant's Global Assessment of Overall Well-being at Week 6/Final Visit.
Description: as for outcome 9
Time Frame: Week 6/Final Visit
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 75 | 83
Participants | 33 | 45
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; The number of participants with at least a 30% improvement in participant's Global Assessment of Overall Well-Being was compared between the two treatment groups using a chi-square test. A 95% CI for the difference in incidence between groups was also computed; Test type: Superiority or Other; p = 0.200, Chi-squared; Mean Difference (Final Values) = -0.102, 95% CI 2-sided [-0.257 to 0.053] — Mean Difference (Final Values) indicates difference in incidence (proportion) between treatments

11. Other Pre Specified Outcome: Change From Baseline in Assessment of Ambulatory Blood Pressure Monitoring (ABPM) for SBP and DBP at Week 6/Final Visit
Description: Ambulatory BP measurements were obtained from 24 participants(in addition to the BP measurements obtained by the cuff technique) participating in the exploratory 24-hour ABPM sub-study. BP was monitored by a 24 hour Ambulatory BP device provided by a central vendor.
Time Frame: 6 weeks/Final Visit
Population: Safety population included all randomized participants who received at least one dose of study medication. For one participant in Naproxen Arm the device failed to collect 11 out of 24 readings at Week 6 and this participant was not included in analysis. ABPM data were analyzed for 12 and 11 participants in Celecoxib and Naproxen Arms respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 12 | 11
mmHg
  SBP | 2.4 (7.02) | -1.7 (12.40)
  DBP | 0.9 (4.23) | -1.1 (5.36)

12. Other Pre Specified Outcome: Change From Baseline in Assessment of ABPM for Heart Rate at Week 6/Final Visit
Description: Ambulatory BP measurements were obtained from 24 participants (in addition to the BP measurements obtained by the cuff technique) participating in the exploratory 24-hour ABPM sub-study. A summary of ABPM 24-hour averages for heart rate is presented in this Outcome Measure.
Time Frame: 6 weeks/Final Visit
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: bpm (beats per minute)
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 12 | 11
bpm (beats per minute) | 2.5 (6.34) | 3.7 (8.50)

13. Other Pre Specified Outcome: Change From Baseline in Assessment of ABPM for SBP and DBP Pressure at Week 6/Final Visit (Sensitivity Analysis Excluding One Participant)
Description: A summary of ABPM 24-hour averages for SBP and DBP are presented in this Outcome Measure. One of the participant in the Naproxen ABPM Arm had clinically implausible high BP values at Baseline. Due to the low number of participants in each Arm (12 and 11) these values had a significant impact on the mean baseline values for the Naproxen Arm. As a result, an additional sensitivity analysis was conducted, excluding this participant (Participant ID 10031002).
Time Frame: 6 weeks/Final Visit
Population: Safety population included all randomized participants who received at least one dose of study medication. A total of 22 out of 24 participants were analyzed in this sensitivity analysis. Two participants were excluded, one due to outlying BP values at Baseline and another due to the device failure to collect 11 out of 24 readings).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 12 | 10
mmHg
  SBP | 2.4 (7.02) | 1.9 (4.13)
  DBP | 0.9 (4.23) | 0.3 (2.86)

14. Other Pre Specified Outcome: Change From Baseline in Assessment of ABPM for Heart Rate at Week 6/Final Visit (Sensitivity Analysis Excluding One Participant)
Description: A summary of ABPM 24-hour averages for heart rate is presented in this Outcome Measure. One of the participant in the Naproxen ABPM Arm had clinically implausible high BP values at Baseline. Due to the low number of participants in each Arm (12 and 11) these values had a significant impact on the mean baseline values for the Naproxen Arm. As a result, an additional sensitivity analysis was conducted, excluding this participant (Participant ID 10031002).
Time Frame: 6 weeks/Final Visit
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Celecoxib | Naproxen
Number analyzed (Participants) | 12 | 10
bpm | 2.5 (6.34) | 3.3 (8.82)

ADVERSE EVENTS:
Time Frame: Up to Week 6/Final Visit
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/98
Other Adverse Events (participants affected / at risk) | 10/100 | 18/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=100) | Naproxen (N=98)
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=100) | Naproxen (N=98)
Nausea (Gastrointestinal disorders) | 4 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Headache (Nervous system disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.